CLINICAL TRIAL: NCT04400591
Title: Expanded Access Protocol (EAP) For Subjects Receiving Lisocabtagene Maraleucel That Is Nonconforming For Commercial Release
Brief Title: Nonconforming Lisocabtagene Maraleucel Expanded Access Protocol
Status: Available | Type: Expanded Access
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: JCAR017-EAP-001; U1111-1251-6894 (Registry Identifier: WHO)
Record Dates: First submitted 2020-05-20; First posted 2020-05-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Expanded Access; JCAR017; Lisocabtagene Maraleucel; CAR T; nonconforming;; relapsed/refractory diffuse large B cell lymphoma; nonconforming lisocabtagene mareleucel; liso-cel
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: Nonconforming Lisocabtagene Maraleucel — Nonconforming lisocabtagene maraleucel is lisocabtagene maraleucel that does not meet the commercial release specifications, however is deemed acceptable to administer as an investigational product in the Expanded Access Protocol setting.
  Other Names: JCAR017

SUMMARY:
This is an expanded access protocol that will be conducted at sites qualified and approved to treat subjects with lisocabtagene maraleucel. Sometimes when lisocabtagene maraleucel is manufactured the drug does not pass all the testing results to be called lisocabtagene maraleucel. When this happens the drug is called nonconforming lisocabtagene maraleucel. The expanded access protocol will be used to allow subjects to receive nonconforming lisocabtagene maraleucel only if the potential benefit is better than the potential risk. This expanded access protocol is restricted to those subjects who were prescribed lisocabtagene maraleucel as part of their routine care.

Subjects will first receive a lymphodepleting chemotherapy regimen and then be treated with nonconforming lisocabtagene maraleucel as the treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. Subject and/or LAR must understand and voluntarily sign an informed consent form prior to any study-related assessments/procedures being conducted.
2. Subject was prescribed lisocabtagene maraleucel (liso-cel) for a diagnosis that is approved per local prescribing information, per treating physician assessment.
3. Subject is ≥ 18 years of age at the time of signing the informed consent form.
4. Subject had a subject-specific batch of liso-cel manufactured intended for commercial treatment; however, the final manufactured product did not meet the local commercial release criteria.
5. Remanufacturing (eg, repeat leukapheresis and manufacturing) is deemed not feasible or clinically inappropriate per assessment of the treating physician in discussion with the subject.
6. Subject is clinically stable, has recovered from any prior toxicities which places the subject at clinical risk prior to receiving LD chemotherapy, and has adequate bone marrow function to receive LD chemotherapy. The treating physician is advised to contact the Medical Monitor in the event there is any concern regarding administration of LD chemotherapy.
7. Females of childbearing potential must:

   1. Have a negative pregnancy test as verified by the treating physician within 7 days prior to the first dose of lymphodepleting chemotherapy following institutional testing methodology practices. This applies even if the subject practices true abstinence from heterosexual contact.
   2. Either commit to true abstinence from heterosexual contact or agree to use, and be able to comply with, effective contraception without interruption. Contraception methods must include 1 highly effective method from screening until at least 12 months after the nonconforming liso-cel administration.
   3. Agree to abstain from breastfeeding during study participation and for at least 12 months following nonconforming liso-cel administration.
   4. There are insufficient exposure data to provide any recommendation concerning the duration of contraception and the abstaining from breastfeeding following treatment with liso-cel. Any decision regarding contraception and breastfeeding after infusion should be discussed with the treating physician.
8. Male subjects must:

   1. Practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential for at least 12 months after nonconforming liso-cel administration even if the subject has undergone a successful vasectomy.
   2. There are insufficient exposure data to provide any recommendation concerning the duration of contraception following treatment with liso-cel. Any decision regarding contraception after infusion should be discussed with the treating physician
9. Subject must agree to not donate blood, organs, tissue, sperm or semen and egg cells for usage in other individuals for at least 1 year following nonconforming liso-cel administration.

Exclusion Criteria:

1. Subject has a hypersensitivity to the active substance or to any of the excipients.
2. Subject should not experience a significant worsening in clinical status that would, in the opinion of the treating physician, either increase the risk of adverse events associated with lymphodepleting chemotherapy, or exclude them from treatment with nonconforming liso-cel.
3. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness, sociologic or geographic condition that would prevent the subject from participating in the Expanded Access Protocol complying with protocol requirements in the Investigator's judgement.
4. Subject has any condition and/or laboratory abnormality that places the subject at unacceptable risk if he/she were to participate in the Expanded Access Protocol based on the Investigator's judgement
5. Pregnant or nursing women or has intention of becoming pregnant during the study.
6. Subjects with primary central nervous system (CNS) lymphoma (note: subjects with secondary CNS involvement are allowed on study).
7. Subject has uncontrolled hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection at the time of pretreatment evaluation
8. Subject has uncontrolled systemic fungal, bacterial, viral or other infection despite appropriate antibiotics or other treatment at the time of nonconforming liso-cel administration.
9. Subject has active acute or chronic graft-versus-host disease (ie, GVHD)
10. Subject should not be actively receiving anticancer treatment that would, in the opinion of the treating physician, either increase the risk of AEs associated with LD chemotherapy or CAR T therapy or interfere with site routine care treatment plan associated with CAR T therapy. The treating physician is advised to consult with the Medical Monitor for case discussion if needed.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html